CLINICAL TRIAL: NCT01010139
Title: A Single Dose, 3-Period, 3-Treatment, 6-Sequence Crossover Pharmacokinetic and Comparative Bioavailability Study of Codeine Sulfate Tablet Formulations Under Fasting Conditions
Brief Title: Pharmacokinetic and Comparative Bioavailability Study of Codeine Sulfate Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CODE-T60-PLFS-1
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O(6)-codeine methyl ether

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Codeine Sulfate — 15 mg, 30 mg and 60 mg Tablet

SUMMARY:
The objective of this study designed to characterize the pharmacokinetics and comparative bioavailability of Roxane Laboratories' codeine sulfate tablets after oral administration of 60 mg doses as 1 x 60 mg, 2 x 30 mg and 4 x 15 mg under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to codeine sulfate or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 21 Days

CONTACTS AND LOCATIONS:
Overall Officials: James P Doherty, DO, Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, San Antonio, Texas, United States